CLINICAL TRIAL: NCT01837966
Title: A Randomized Prospective Placebo-Controlled Study of the Effects of Lavender Aromatherapy on Preoperative Anxiety in Breast Surgery Patients
Brief Title: Randomized, Placebo-Controlled Study: Effects of Lavender Aromatherapy on Preoperative Anxiety in Breast Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03152
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Anxiety; Generalized; Breast Diseases; Surgery
Keywords: re-operative anxiety; breast surgery; lavender oil; aromatherapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Breast Diseases | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lavender oil (Active Comparator): Lavender oil aromatherapy
  Interventions: Other: Lavender oil
- Placebo (Placebo Comparator): Placebo -- unscented oil aromatherapy
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lavender oil — 2 drops for aromatherapy
  Arms: Lavender oil
Other: Placebo — 2 drops unscented mineral oil for aromatherapy
  Arms: Placebo

SUMMARY:
The study is designed to see if lavender aroma therapy reduces pre-operative anxiety in breast surgery patients.

DETAILED DESCRIPTION:
Many patients undergoing surgery experience anxiety in the preoperative setting. Pharmacologic anxiolytics require monitoring and cause excess sedation which often interferes with the ability to assess and obtain consent from a patient in the preoperative holding area. Lavender aromatherapy is an alternative treatment for anxiety which is safe, inexpensive, easy to administer, and not overly sedating. In addition to its benefits in the preoperative setting, anxiolysis and reduction in sympathetic drive can lead to reduction in the intraoperative anesthetic and postoperative analgesic requirements. This in turn can lead to faster recovery and expedited discharge from the post anesthesia care unit.

In the proposed study, we would evaluate the efficacy of aromatherapy with lavender oil in reducing anxiety prior to breast surgery. The study group would receive lavender oil preoperatively and the placebo group would receive unscented oil preoperatively. Before and after treatment, anxiety level would be measured using the Spielberger State-Trait Anxiety Inventory. Additionally, vital signs and Bispectral index (BIS) will be measured before and after treatment, as further indicators of anxiety level. We hypothesize that lavender aromatherapy will decrease anxiety and subsequently will reduce blood pressure, heart rate, and BIS.

ELIGIBILITY:
Inclusion Criteria: Female; Age 18+; American Society of Anesthesiologists (ASA) I-III; undergoing elective breast surgery

Exclusion Criteria: Male; History of asthma/bronchitis/Chronic Obstructive Pulmonary Disease (COPD)/contact dermatitis to cosmetic fragrances/pregnancy; significant laboratory abnormalities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wajda, MD, Study Director — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kil HK, Kim WO, Chung WY, Kim GH, Seo H, Hong JY. Preoperative anxiety and pain sensitivity are independent predictors of propofol and sevoflurane requirements in general anaesthesia. Br J Anaesth. 2012 Jan;108(1):119-25. doi: 10.1093/bja/aer305. Epub 2011 Nov 13. PMID 22084330
- [Background] Nelson JP, Glassburn AR Jr, Talbott RD, McElhinney JP. Horizontal flow clean room. Bacteriologic studies. Rocky Mt Med J. 1975 Jun;72(6):243-6. No abstract available. PMID 1096279
- [Background] Moss M, Cook J, Wesnes K, Duckett P. Aromas of rosemary and lavender essential oils differentially affect cognition and mood in healthy adults. Int J Neurosci. 2003 Jan;113(1):15-38. doi: 10.1080/00207450390161903. PMID 12690999
- [Background] Barocelli E, Calcina F, Chiavarini M, Impicciatore M, Bruni R, Bianchi A, Ballabeni V. Antinociceptive and gastroprotective effects of inhaled and orally administered Lavandula hybrida Reverchon "Grosso" essential oil. Life Sci. 2004 Nov 26;76(2):213-23. doi: 10.1016/j.lfs.2004.08.008. PMID 15519366
- [Background] Kim S, Kim HJ, Yeo JS, Hong SJ, Lee JM, Jeon Y. The effect of lavender oil on stress, bispectral index values, and needle insertion pain in volunteers. J Altern Complement Med. 2011 Sep;17(9):823-6. doi: 10.1089/acm.2010.0644. Epub 2011 Aug 19. PMID 21854199
- [Background] Orbach-Zinger S, Ginosar Y, Elliston J, Fadon C, Abu-Lil M, Raz A, Goshen-Gottstein Y, Eidelman LA. Influence of preoperative anxiety on hypotension after spinal anaesthesia in women undergoing Caesarean delivery. Br J Anaesth. 2012 Dec;109(6):943-9. doi: 10.1093/bja/aes313. Epub 2012 Sep 10. PMID 22964265
- [Background] Oliphant SS, Lowder JL, Ghetti C, Zyczynski HM. Effect of a preoperative self-catheterization video on anxiety: a randomized controlled trial. Int Urogynecol J. 2013 Mar;24(3):419-24. doi: 10.1007/s00192-012-1868-y. Epub 2012 Jul 3. PMID 22752014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the out-patient surgical unit of New York University (NYU) Langone Medical Center from January 18 - June 11, 2013. Only female patients having breast surgery were approached.
Pre-assignment Details: Only patients who had any allergy or sensitivity to the oils or had allergies were excluded.
Period: Overall Study
Arm/Group | Lavender Oil | Placebo
Started | 47 | 46
Completed | 45 | 45
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: 93 patients were enrolled into the study, but only 88 had useable data. 43 patients in the lavender arm and 45 in the placebo/unscented oil arm had usable data.
Groups:
- Placebo: Placebo - unscented oil aromatherapy
  Placebo: 2 drops unscented mineral oil for aromatherapy
- Total: Total of all reporting groups
Arm/Group | Lavender Oil | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Continuous [Mean (Full Range); unit: years] | 50 [24 to 86] | 48 [22 to 82] | 49 [22 to 86]
Sex/Gender, Customized [Number; unit: participants]
  Male | 0 | 0 | 0
  Female | 43 | 45 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13
American Society of Anesthesiologists (ASA) Physical Status Classification [Number; unit: participants] — ASA Physical Status I, II, III
  ASA I: Normal healthy patient (excludes the very young/very old) ASA II - Patients w/ mild systemic disease (No functional limitations; well-controlled disease of one body system; i.e. controlled HTN or diabetes w/o systemic effects, cigarette smoking w/o COPD) ASA III - Patients w/ severe systemic disease (Some functional limitation; controlled disease of more than one body system/or one major system; no immediate danger of death; i.e controlled Congestive Heart Failure, stable angina, old heart attack, poorly controlled HTN)
  participants
    ASA I | 15 | 15 | 30
    ASA II | 27 | 29 | 56
    ASA III | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Reduction
Description: We hoped to show that lavender aroma therapy reduces preoperative anxiety in patients undergoing breast. The Trait subscale (STAI-TRAID) of the Spielberger State-Trait Anxiety Inventory was administered before and after 10 minutes of aromatherapy treatment pre-surgery. The TRAIT subscale contains 20 questions scored on a Likert scale from 1-4; item scores are summed for a total score ranging from 20 to 80, with higher scores indicating higher anxiety. Change in anxiety was calculated as the score pre-aromatherapy minus the score post-aromatherapy. Higher positive change scores indicate greater reductions in anxiety.
Time Frame: 20 minutes before surgery (pre aromatherapy) and 10 minutes before surgery (post aromatherapy)
Population: Analysis of STAI-TRAIT questions
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lavender Oil: Lavender oil aromatherapy
  Lavender oil: 2 drops for aromatherapy
  There were no adverse events for this arm.
- Placebo: Placebo -- unscented oil aromatherapy
  Placebo: 2 drops unscented mineral oil for aromatherapy
  There were no adverse events for this arm.
Arm/Group | Lavender Oil | Placebo
Number analyzed (Participants) | 43 | 45
units on a scale | 0.89 (.32) | .74 (.44)

ADVERSE EVENTS:
Arm/Group | Lavender Oil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 0/43 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No